CLINICAL TRIAL: NCT00351858
Title: Phase II Study of the Trifunctional Anti-HER-2/Neu x Anti-CD3 Antibody Ertumaxomab for Hormone Therapy Refractory Patients With Her-2/Neu 1+ or 2+ Expressing Advanced or Metastatic Breast Cancer
Brief Title: Safety and Efficacy Study of the Trifunctional Antibody Ertumaxomab to Treat Patients With Advanced or Metastatic Breast Cancer
Acronym: IV REXBC 02
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: company focus on other projects
Sponsor: Neovii Biotech (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBT-IVREXBC 02; EudraT number: 2005-004294-21
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast Cancer; investigational drug; drug therapy; Antineoplastic Protocols; Immunotherapy; Metastatic breast cancer; Advanced breast cancer; Stage III to IV breast cancer; Hormonal therapy refractory; Failure of hormonal therapy; Her-2/neu expressing breast cancer; low to moderate Her-2/neu expression
MeSH Terms: conditions — Breast Neoplasms | interventions — ertumaxomab

INTERVENTIONS:
Drug: ertumaxomab

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the investigational trifunctional anti-Her-2/neu x anti-CD3 antibody ertumaxomab as treatment for hormone therapy refractory Her-2/neu 1+ or 2+ expressing advanced or metastatic breast cancer

DETAILED DESCRIPTION:
A multi-centre, phase II study of ertumaxomab in metastatic breast cancer patients who became progressive after hormonal therapy. Each eligible patient will receive three ascending doses of ertumaxomab, administered intravenously. Ertumaxomab will be administered as a 3-hour constant rate infusion with a dosing interval of 7 days. Each patient will participate in this study for up to 7 months (includes the up to 21 days screening period, 14 days treatment period, and up to 180 days/6 months follow-up), with 3-monthly post-study follow-up until the patient becomes progressive.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, and if of child-bearing potential must have negative pregnancy test result within 2 days before enrolment and must agree to practice effective birth control during the study.
* Aged 18 years and older.
* Histologically or cytologically confirmed invasive breast cancer with stage IIIb or IV disease with documented progression.
* Measurable disease according to RECIST.
* Histologically documented advanced primary breast cancer or biopsy of metastatic site demonstrating HER-2/neu expression (HER-2/neu 1+ or 2+, determined by immunohistochemistry [IHC]). HER-2/neu 2+ patients must have a negative Fluorescence In Situ Hybridization [FISH] test result.
* Hormone receptor status Estrogen Receptors (ERs) positive and/or Progesterone Receptors (PRs) positive.
* No prior treatment with mouse or rat antibodies.
* Life expectancy of at least six months (if the life expectancy of a patient is unspecified she will be allowed to enter the study).
* An Eastern Cooperative Oncology Group (ECOG) performance score of £ 1.
* Patients must have had disease progression after hormonal therapy including at least one aromatase inhibitor.
* Adequate hematological, liver and kidney function:

  * Thrombocytes ³ 100000 / mm³ (= 100 x 109 /l)
  * Hemoglobin ³ 10 g/dl
  * Neutrophil count ³ 1500/mm³ (= 1.5 x 109 /l)
  * WBC ³ 3 X 109 /l
  * Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) ≤ 2.5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 2 x ULN
  * Creatinine ≤ 1.5 x ULN or clearance ³ 60 ml/min
* No life-threatening visceral disease.
* No known brain or central nervous system metastases.
* No symptomatic pleural effusions.
* No symptomatic pericardial effusions.
* No subjects whose only site of metastatic involvement is bone metastases with the exception of those with a measurable soft tissue component of the bone lesion seen with imaging that does not require palliative radiation intervention and/or the patient has a lytic bone lesion ³ 1 cm measured with radiography that can be followed for evidence of re-calcification.
* No history of relevant cardiovascular disease:

  * LVEF within the institutional ranges of normal as measured by echocardiogram or MUGA scan
  * No prior uncontrolled or symptomatic congestive heart failure NYHA ³ 2
  * No myocardial infarction within the past two years
  * No uncontrolled or symptomatic cardiac arrhythmias
* No severe dyspnea.
* No pulmonary dysfunction or need for continuous supportive oxygen inhalation.
* No other concurrent uncontrolled co-morbid illness.
* No other concurrent malignancy, except treated basal cell or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix.
* Patients with documented autoimmune diseases (such as lupus) are excluded from participation in the study unless a waiver is granted by the responsible medical monitor.
* Patients with a human immunodeficiency virus, hepatitis B or hepatitis C positive status are excluded from participation in the study.
* No prior or concurrent chemotherapy regimen for advanced or metastatic disease.
* Prior neo-adjuvant or adjuvant chemotherapy is allowed provided it was stopped at least six months before study entry.
* No concurrent hormone therapy (hormone therapy must be stopped at the screening visit).
* At least 4 weeks since prior radiotherapy.
* No concurrent immune therapy.
* No concurrent corticosteroid therapy.
* No regularly used medication for a health condition or comorbidity that might result in undue risk to the patient.
* No prior investigational treatment for advanced or metastatic disease.
* Able and willing to comply fully with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate clinical efficacy of the investigational trifunctional antibody ertumaxomab for the treatment of hormone therapy refractory advanced or metastatic breast cancer tumors (stage IIIb or IV) which are known to express Her-2/neu (1+ or 2+)

SECONDARY OUTCOMES:
Time to progression
Duration of response
Time to response
Clinical benefit of ertumaxomab (defined as the rate of confirmed complete remission, partial remission and stable disease)
Tumor marker levels (CA 15-3 and CEA)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Cardoso, MD, Principal Investigator — Brussels
Locations (1):
- Jules Bordet Institute, Free University of Brussels, Brussels, Belgium

REFERENCES:
- [Background] Kiewe P, Hasmuller S, Kahlert S, Heinrigs M, Rack B, Marme A, Korfel A, Jager M, Lindhofer H, Sommer H, Thiel E, Untch M. Phase I trial of the trifunctional anti-HER2 x anti-CD3 antibody ertumaxomab in metastatic breast cancer. Clin Cancer Res. 2006 May 15;12(10):3085-91. doi: 10.1158/1078-0432.CCR-05-2436. PMID 16707606
- [Background] Lindhofer H, Mocikat R, Steipe B, Thierfelder S. Preferential species-restricted heavy/light chain pairing in rat/mouse quadromas. Implications for a single-step purification of bispecific antibodies. J Immunol. 1995 Jul 1;155(1):219-25. PMID 7602098
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Zeidler R, Mayer A, Gires O, Schmitt B, Mack B, Lindhofer H, Wollenberg B, Walz A. TNFalpha contributes to the antitumor activity of a bispecific, trifunctional antibody. Anticancer Res. 2001 Sep-Oct;21(5):3499-503. PMID 11848515